CLINICAL TRIAL: NCT01931930
Title: Effect of Perilla Extract on Improvement of Intestinal Discomfort and Bowel Function in Healthy Volunteers With Gastrointestinal Discomfort
Brief Title: Effect of Perilla Extract on Improvement on Gastrointestinal Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amino Up Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BTS656/12
Record Dates: First submitted 2013-08-23; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Abdominal Pain/ Discomfort; Slightly Constipation
Keywords: Gastrointestinal discomfort; Perilla frutescens; bloating; abdominal discomfort; human study; healthy subjects
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perilla extract (Experimental): Experimental arm: Perilla extract
  Interventions: Dietary Supplement: Perilla extract
- Maltodextrin (Placebo Comparator): Placebo arm: Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Perilla extract
  Arms: Perilla extract
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
In the current study the effects of proprietary Perilla frutescens leaf extract in comparison to Maltodextrin, a fully digestible carbohydrate (placebo control), on gastrointestinal discomfort and bowel function were investigated. The study was performed double-blind and placebo-controlled with a 4 week intervention period. Study products were taken two times daily (each one capsule before breakfast and dinner).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without clinical diagnosed diseases with relevant effect on the gastrointestinal system or on visceral motility.
* BMI: 19-30 kg/m2
* Reduced bowel movements defined as an average of >1 and ≤ 3.5 stools per week for at least the previous 6 months
* Gastrointestinal symptoms of at least 5 points
* Male or female
* Age ≥ 30 and ≤ 70 years
* Nonsmoker
* Written consent to participate in the study
* Able and willing to follow the study protocol procedures

Exclusion Criteria:

* Subject under prescription for medication for digestive symptoms such as anti-spasmodic, laxatives and anti-diarrheic drugs or other digestive auxiliaries
* Relevant history, presence of any medical disorder or intake of medication / dietary supplements, potentially interfering with this trial at screening
* Subjects with stool frequency of ≤ 1 stool every 7 days or > 3,5 stools per week
* Subjects not willing to avoid pre- and probiotics for the duration of the study
* Intake of antibiotics in the last 4 weeks and laxatives in the last 2 weeks
* Change of dietary habits within the 4 weeks prior to screening (for instance start of a diet high in fibers)
* Pregnant subject or subject planning to become pregnant during the study; breast-feeding subject.
* Subjects with history of drug, alcohol or other substances abuse, or other factors limiting their ability to co-operate during the study.
* Participants anticipating a change in their lifestyle or physical activity levels since this may also influence the results.
* Known food intolerance or allergy.
* Subject involved in any clinical or food study within the preceding month

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
daily gastrointestinal symptoms | was assessed daily during 4 week intervention
  The following gastrointestinal were rated and reported by the study participants on a daily based. Bloating, rumbling, feeling of fullness, passage of gas, abdominal discomfort (pain and cramps). The rating was done based on a number scale. 0 not at all and 4 extremely.

SECONDARY OUTCOMES:
validated questionnaires | assessed at visit 1 (before) and at visit 2 (after 4 week intervention)
  Three validated questionnaires were used. Two of them were specially designed to evaluate gastrointestinal symptoms and quality of life of people with constipation. The third questionnaire was a validated questionnaire to report stress levels and related changes of stress levels.
  1. Patient assessment of constipation symptoms (PAC SYM)
  2. Patents assessment of constipation quality of life (PAC QOL)
  3. Perceived stress questionnaire (PSQ20)
stool consistency | reported at days with stool during 4 week intervention
  The stool consistency was rated referring to the Bristol stool scale. A scale indicated with pictures how the stool consistency can be rated.
Adverse events | assessed at visit 1 (before) and at visit 2 (after 4 week intervention)
  All adverse events which might be linked to the study product were reported. As the tested study product is a food product being safe for consumption as food no specific parameter to define safety were defined.
Stool frequency | reported at days with stool during 4 week intervention
  The stool frequency was reported on each day with bowel movement.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, PhD, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

REFERENCES:
- [Derived] Buchwald-Werner S, Fujii H, Reule C, Schoen C. Perilla extract improves gastrointestinal discomfort in a randomized placebo controlled double blind human pilot study. BMC Complement Altern Med. 2014 May 27;14:173. doi: 10.1186/1472-6882-14-173. PMID 24885816